CLINICAL TRIAL: NCT05406739
Title: Physiological and Behavioral Regulation of Feeding After Spinal Cord Injury
Brief Title: Feeding Regulation in SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Gary Farkas, Postdoctoral Associate, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20220407
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injuries
Keywords: gut; eating; appetite; hormone
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Cord Injury Group (Experimental): Participants who have a spinal cord injury will receive two meals on two separate visits between five to seven days.
  Interventions: Other: Test Meals
- Control Group (Active Comparator): Participants without a spinal cord injury will receive two meals on two separate visits between five to seven days.
  Interventions: Other: Test Meals

INTERVENTIONS:
Other: Test Meals — For the first meal, Participants will be fasted for 8 hours and will consume a test meal of 255 calories (120 g egg substitute [60 kcal]; 2 slices of bread [120 kcal] with 30 g strawberry jam [75 kcal]; 72% carbohydrate, 24% protein, 2% fat, and 2% fiber) with 120 mL of water.
  After five to seven days, participants will be fasted for 10 hours and will consume a second test meal of 510 calories (240 g egg substitute [120 kcal]; 4 slices of bread [240 kcal] with 60 g strawberry jam [150 kcal]; 72% carbohydrate, 24% protein, 2% fat, and 2% fiber) with 240 mL of water.

SUMMARY:
The overall purpose of this research is to understand the reasons why persons with spinal cord injuries eat more calories than they need to "burn", stay alive, and function. This research will investigate how quickly food moves through a participant's body, the hormones in the participant's body that control energy and digestion, and a participant's impressions of hunger after eating a meal. This will be compared in persons with and without a spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injury (SCI) Participants:

1. Adults (≥ 18 years) with tetraplegia (C5-C8) or paraplegia (T1-L2) SCI
2. Chronic SCI, denoted as ≥ 12 months post-injury
3. American Spinal Injury Association Impairment Scale164 A, B, and C
4. Persons with tetraplegia self-report they are able to feed themselves
5. Self-report on a bowel care program every-other-day
6. English speaking

Control Group (Healthy) Participants:

1. Adults (≥ 18 years) without a SCI (will be sex- and age-matched to persons with SCI)
2. English speaking

Exclusion Criteria:

For All Participants:

1. Currently on a weight loss program/diet and/or actively trying to lose weight
2. Have a self-reported history of

   * Diabetes
   * Thyroid disease
   * Gastrointestinal disease
   * Previous abdominal surgery ≤ 3 months prior to the study
   * Peripheral nervous system prosthesis
   * Swallowing disorders
3. Self-reported food allergies to or dislike the test meals.
4. Self-reported use of a prokinetic agent, antipsychotic agent, or Glucagon like Peptide 1 (GLP-1) agonists
5. Individuals who are not yet adults (infants, children, teenagers)
6. Women that self-report they are pregnant or likely to become pregnant
7. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | Up to seven days
  Gastric emptying will be measured by the SmartPill Wireless Motility Capsule
Upper gastrointestinal transit time | Up to seven days
  Upper gastrointestinal transit time will be measured by the SmartPill Wireless Motility Capsule

SECONDARY OUTCOMES:
Change in postprandial ghrelin | Before the second test meal (up to 7 days) and up to 120 minutes after the second test meal (up to 7 days).
  Measured by serum blood samples
Change in postprandial peptide tyrosine tyrosine (PYY) | Before the second test meal (up to 7 days) and up to 120 minutes after the second test meal (up to 7 days).
  Measured by serum blood samples
Change in postprandial cholecystokinin (CKK) | Before the second test meal (up to 7 days) and up to 120 minutes after the second test meal (up to 7 days).
  Measured by serum blood samples
Change in postprandial Glucagon Peptide 1 (GLP-1) | Before the second test meal (up to 7 days) and up to 120 minutes after the second test meal (up to 7 days).
  Measured by serum blood samples
Change in subjective appetite rating as measured by Palatability Series Visual Analogue Scale | Baseline and up to 7 days
  Change in subjective appetite rating will be measured by Palatability Series Visual Analogue Scale that ranges from 0 mm as "not pleasant" to 100 mm as "extremely pleasant"
Change in subjective appetite rating as measured by Hunger Series Visual Analogue Scale | Baseline and up to 7 days
  Change in subjective appetite rating will be measured by Hunger Series Visual Analogue Scale that ranges from 0 mm as "not at all hungry" to 100 mm as "totally/a lot/very hungry".
Total percentage body fat | Baseline
  Measured by Dual x-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Farkas, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farkas GJ, Sneij A, McMillan DW, Tiozzo E, Nash MS, Gater DR Jr. Energy expenditure and nutrient intake after spinal cord injury: a comprehensive review and practical recommendations. Br J Nutr. 2022 Sep 14;128(5):863-887. doi: 10.1017/S0007114521003822. Epub 2021 Sep 23. PMID 34551839
- [Background] Farkas GJ, Sneij A, Gater DR Jr. Dietetics After Spinal Cord Injury: Current Evidence and Future Perspectives. Top Spinal Cord Inj Rehabil. 2021;27(1):100-108. doi: 10.46292/sci20-00031. PMID 33814888
- [Background] Farkas GJ, Sneij A, Gater DR Jr. Energy Expenditure Following Spinal Cord Injury: A Delicate Balance. Top Spinal Cord Inj Rehabil. 2021;27(1):92-99. doi: 10.46292/sci20-00030. PMID 33814887
- [Background] Farkas GJ, Gater DR. Energy Expenditure and Nutrition in Neurogenic Obesity following Spinal Cord Injury. J Phys Med Rehabil. 2020;2(1):11-13. No abstract available. PMID 32226945
- [Background] Farkas GJ, Pitot MA, Gater Jr. DR. A Systematic Review of the Accuracy of Estimated and Measured Resting Metabolic Rate in Chronic Spinal Cord Injury. Int J Sport Nutr Exerc Metab. 2019 Sep 1;29(5):548-558. doi: 10.1123/ijsnem.2018-0242. PMID 31034249
- [Background] Farkas GJ, Gorgey AS, Dolbow DR, Berg AS, Gater DR. Caloric Intake Relative to Total Daily Energy Expenditure Using a Spinal Cord Injury-Specific Correction Factor: An Analysis by Level of Injury. Am J Phys Med Rehabil. 2019 Nov;98(11):947-952. doi: 10.1097/PHM.0000000000001166. PMID 30817378
- [Result] Farkas GJ, Pitot MA, Berg AS, Gater DR. Nutritional status in chronic spinal cord injury: a systematic review and meta-analysis. Spinal Cord. 2019 Jan;57(1):3-17. doi: 10.1038/s41393-018-0218-4. Epub 2018 Nov 12. PMID 30420688